CLINICAL TRIAL: NCT06830291
Title: Validation and Standardisation of a "Neuralix" Digital Ecological Battery
Acronym: VANOLIX
Status: Recruiting | Type: Observational
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2019PPRC08; 2023-A01562-43 (Other: ANSM IDRCB)
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-03

CONDITIONS: Traumatic Brain Injuries
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- G1 : Control group: single assessment: healthy volunteers undergo the test battery only once
- G2 :Control group: double assessment: healthy volunteers undergo the test battery twice, six months apart
- G3 :Patient group: single assessment: patients undergo the test battery only once
- G4 : Patient group: double assessment: patients undergo the test battery twice, six months apart

SUMMARY:
The management of head trauma patients requires the assessment of cognitive disorders using standardized neuropsychological tests and questionnaires. However, the evaluation tools currently available present well-identified limitations limiting the accuracy of the measurements (in a non-exhaustive manner, let us cite for example the absence of control of the rate of "false positives" or even the impossibility of measuring the improvement or decline in performance over time). In order to overcome these limitations, the Neuralix battery was created with particular attention to the assessment of memory and executive functions largely impacted after head trauma. The Neuralix battery comes in the form of a digital application accessible online and allowing a global assessment of cognitive functions in adults. In addition, the processing of results includes the operationalization of decision criteria taking into account the limitations cited above in order to improve the sensitivity of the evaluation.

The VANOLIX study proposes the validation of the Neuralix cognitive battery with head trauma patients of moderate to severe intensity as well as its standardization with healthy volunteers, these two steps being essential to making the tool available to clinician-researchers.

ELIGIBILITY:
Inclusion Criteria:

* French-speaking subject aged 18 to 65 years old
* Signed consent to participate
* History of head trauma of moderate to severe intensity, i.e. having presented the high risk criteria of the study by Masters et al. (1987) at the time of the head trauma, and occurred a maximum of 5 years after inclusion in the VANOLIX study

Exclusion Criteria:

* Visual or hearing or motor deficit disrupting the taking of cognitive tests
* Subject with insufficient knowledge of counting (up to 25), the alphabet, reading, or French writing
* Subject with a severe intellectual disability
* Subject with past psychiatric or behavioral disorders requiring a stay >2 days in a specialized environment or requiring current treatment other than a single anxiolytic
* Current treatment with antidepressant
* Current treatment with antipsychotic or multiple anxiolytics
* Single anxiolytic treatment initiated or increased for less than 1 month or current antiepileptic treatment
* Subject with a neurological condition or a history leading to cerebral dysfunction likely to interfere with the cognitive assessment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with TBI moderate to severe vs controls
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Sensitivity og the Neuralix Battery | 36 month
  Determine the sensitivity of the Neuralix battery to cognitive disorders post-head trauma of moderate to severe intensity.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital d'Instruction des Armées - Percy, Clamart, France